CLINICAL TRIAL: NCT03140072
Title: A Phase I, Randomized, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Single and Multiple Ascending Oral Doses of AZD9898 in Healthy Volunteers and Asthma Patients.
Brief Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of AZD9898
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated based on interim review
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7620C00001
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: Asthma, Single Ascending Dose (SAD), Multiple Ascending Dose (MAD), AZD9898
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD9898 (Experimental): In Part 1 of the study, 5 single dose cohorts are planned to be evaluated, where AZD9898 will be administered. Eight subjects will participate in each cohort. Within each cohort, 6 (alternatively 8 or 10) subjects will be randomized to receive a single dose of AZD9898. Fifteen asthma patients are planned to participate in 3 cohorts in Part 2. Five patients will participate in each cohort. Within each cohort, 4 (alternatively 6 or 8) patients will be randomized to receive a single dose of AZD9898. In Part 3, 3 dose cohorts are planned. Nine healthy subjects will participate in each cohort. Within each cohort, 6 (alternatively 8, 10 or 12) subjects will be randomized to receive AZD9898. The subjects taking part in one of the MAD cohorts under fasted conditions will also take part in Part 3B in order to explore the influence of food on the PK of AZD9898.
  Interventions: Drug: AZD9898
- Placebo (Placebo Comparator): In Part 1 of the study, 5 single dose cohorts are planned to be evaluated, where matching placebo will be administered. Eight subjects will participate in each cohort. Within each cohort, 2 (alternatively 3) subjects will be randomized to receive a single dose of matching placebo. Fifteen asthma patients are planned to participate in 3 cohorts in Part 2. Five patients will participate in each cohort. Within each cohort, one patient (alternatively 2 or 3 patients) will be randomized to receive a single dose of matching placebo. In Part 3, 3 dose cohorts are planned. Nine healthy subjects will participate in each cohort. Within each cohort, 3 (alternatively 4) subjects will be randomized to receive matching placebo.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: AZD9898 — In Parts 1 and 2 of the study, each subject/patient will receive a single dose (one dose level) of AZD9898, under fasted conditions. Starting dose in part 1 (SAD in healthy subjects) is 3 mg, subsequent doses will be selected based on emerging data. In Part 3 of the study, each subject will receive one dose level of AZD9898, once daily, under fasted or fed conditions. Subjects participating in Part 3B (food effect cohort) will receive an additional administration of the same dose, on the last day to investigate the effects of food.
  Arms: AZD9898
Drug: Matching Placebo — In Parts 1 and 2 of the study, each subject/patient will receive a single dose (one dose level) of matching placebo, under fasted conditions. In Part 3 of the study, each subject will receive one dose level of matching placebo, once daily, under fasted or fed conditions. Subjects participating in Part 3B (food effect cohort) will receive an additional administration of the same dose, on the last day to investigate the effects of food.
  Arms: Placebo

SUMMARY:
In this integrated, multi-part, Phase I study, the safety, tolerability, food effect, pharmacokinetic (PK) and pharmacodynamic (PD) properties of single and repeated doses of AZD9898 will be investigated.

DETAILED DESCRIPTION:
This study will be a Phase I, randomized, placebo-controlled study in healthy subjects and asthma patients, performed at 2 study centers. The study will consist of 3 parts (Part 1 [SAD in healthy subjects]; Part 2 [SAD in asthma patients]; Part 3 [MAD in healthy subjects under fasted conditions, with one cohort participating under fed conditions during one day as well]). The SAD cohorts in Parts 1 and 2 of the study will include male and women of non-childbearing potential (WONCBP) until the exposure limit for males has been reached. If an additional cohort for Parts 1 and 2 with a dose exceeding exposure limits in males is warranted (to explore the upper end of the dose response curve), this will be conducted in WONCBP only. Cohorts in Part 3 will include male subjects and WONCBP, depending on recruitment feasibility. All cohorts in the study will be single-blinded.

ELIGIBILITY:
Inclusion Criteria:

* For Parts 1 and 3:

  * Healthy male and female subjects aged 18 to 50 years.
  * All females must have a negative pregnancy test at the screening visit and on admission to the clinical unit, must not be lactating and must be of non-childbearing potential. • Has a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

For Part 2:

* In addition to the inclusion criteria for Parts 1 and 3, Male and female subjects aged 18 to 60 years.
* Has been diagnosed by a physician with asthma for at least 12 months prior to the screening visit.
* Has an FEV1 ≥ 65% at the screening visit and prior to dosing on Day 1, as measured before administration of a bronchodilator at both time points.
* Has been on stable standard asthma treatment.

Exclusion Criteria:

* For Parts 1,2,3:

  * History of any clinically important disease or disorder.
  * History of unstable psychiatric disorders.
  * History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with the drugs.
  * Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the screening visit or the first administration of IMP.
  * Any clinically important abnormalities in hematology, clinical chemistry or urinalysis results at the screening visit or on admission.
  * Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV) type I and II antibodies.
  * Abnormal vital signs. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG.
  * Prolonged QTcF > 450 ms or shortened QTcF < 340 ms.
  * PR (PQ) interval shortening. PR (PQ) interval prolongation.
  * Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms.
  * Subjects with QRS > 110 ms, but < 115 ms are acceptable if there is no evidence of, e.g., ventricular hypertrophy or pre-excitation.
  * Known or suspected history of drug abuse.
  * Current smokers or those who have smoked or used nicotine products within the previous 3 months.
  * History of alcohol abuse.
  * Positive testing for drugs of abuse or alcohol or cotinine at the screening visit or on admission.
  * History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
  * Excessive intake of caffeine-containing drinks or food.
  * Use of drugs with enzyme inducing properties.
  * Apart from use of required asthma medication, use of any other prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
  * Use of any prescribed or non-prescribed leukotriene modifiers (e.g., montelukast) within 3 months prior to administration of IMP.
  * Hormone replacement therapy is not allowed for females, in order to exclude any drug-drug interaction.
  * Plasma donation within one month of the screening visit or any blood donation/blood loss exceeding 500 mL during the 3 months prior to the screening visit.
  * Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study.
  * Subjects who have previously received AZD9898.
  * Involvement of any AstraZeneca or study center employee or their close relatives.
  * Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data.
  * Subjects who are vegans or have medical dietary restrictions (only applicable for volunteers participating in the food effect cohort in Part 3 of the study).
  * Subjects who cannot communicate reliably with the Investigator.
  * Vulnerable subjects.
  * Male subjects with a female partner already pregnant at the time of the screening visit will be excluded from the study.
  * Previous bone marrow transplant. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

For part 2:

* If SABAs are used, serum or plasma potassium levels must be within the normal range and not lower than 3.8 mEq/L at the screening visit and on admission.
* Meet any of the standard Hy's Law criteria at the screening visit or on admission.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) | Change from baseline up to follow-up (7-10 days after last dose)
  To assess the adverse events as a criteria of safety and tolerability variables.
Vital sign (Blood pressure [BP]) | Change from baseline up to follow-up (7-10 days after last dose)
  To assess the vital signs as a criteria of safety and tolerability variables.
Vital sign (pulse) | Change from baseline up to follow-up (7-10 days after last dose)
  To assess the vital sign as a criteria of safety and tolerability variables.
Vital sign (temperature) | Change from baseline up to follow-up (7-10 days after last dose)
  To assess the vital sign as a criteria of safety and tolerability variables.
Resting and digital electrocardiograms (ECGs) | Change from baseline up to follow-up (7-10 days after last dose)
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Cardiac telemetry | Change from baseline up to Post-dose (at least 30 minutes pre-dose until at least 24 hours post-dose)
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Physical examination | Change from baseline up to follow-up (7-10 days after last dose)
  To assess the physical conditions as a criteria of safety and tolerability variables.
Laboratory assessments (hematology, clinical chemistry and urinalysis) | Change from baseline up to follow-up (7-10 days after last dose)
  To assess hematology, clinical chemistry and urinalysis as a criteria of safety and tolerability variables.

SECONDARY OUTCOMES:
PK assessment: Cmax (Observed maximum plasma concentration taken directly from the individual concentration-time curve) | Parts 1,2: Days 1,2,3, For Part 3: Days 1, 2, 3,4, 5, 6 and up to Day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: Ctrough (Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration])) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: tmax (Time to reach maximum plasma concentration, taken directly from the individual concentration-time curve) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: λz (Terminal rate constant, estimated by log-linear least-squares regression of the terminal part of the concentration-time curve) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: t1/2λz (Terminal half-life, estimated as (ln2)/λz) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: tlast (Time of last quantifiable plasma concentration) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: AUC(0-last) (Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration, calculated by linear up/log down trapezoidal summation) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: AUC (Area under the concentration-time curve in the plasma from zero (pre-dose) extrapolated to infinite time) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: AUC(0-12) (Area under the plasma concentration-curve from time zero to 12 hours post-dose) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: AUC(0-24) (Area under the plasma concentration-curve from time zero to 24 hours post-dose) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: CL/F (Apparent oral clearance estimated as dose divided by AUC) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: CLss/F (Apparent oral clearance at steady state) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: MRT (Mean residence time) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: Vz/F (Apparent volume of distribution during terminal phase (extravascular administration)) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: Vss/F (Apparent volume of distribution at steady state (extravascular administration)) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: AUC(0-24)/D (Dose normalized AUC(0-24), estimated by dividing AUC(0-24) by the dose administered) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: AUC/D (Dose normalized AUC, estimated by dividing AUC by the dose administered) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: Cmax/D (Dose normalized Cmax, estimated by dividing Cmax by the dose administered) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: Rac (Accumulation ratio) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PK assessment: TCP (Time change parameter) | Parts 1,2: At days 1,2,3, For Part 3: At days 1, 2, 3,4, 5, 6 and up to day 12 as needed, 7-13 days post first dose, 8-14 days post first dose
  Evaluation of the PK of AZD9898 in Parts 1 (single ascending dose in healthy subjects), 2 (single ascending dose in asthma patients) and 3 (multiple ascending dose in healthy subjects) and multiple dose IMP administration under fed and fasted conditions in Part 3 of the study.
PD Parameter: Plasma 4-β-hydroxy-cholesterol (Part 3 only) | Day -1 and last dosing day
  The plasma 4-β-hydroxy-cholesterol at baseline versus after treatment will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, Principal Investigator — PAREXEL Early Phase Clinical Unit London; Dave Singh, Principal Investigator — The Medicines Evaluation Unit
Locations (2):
- United Kingdom (2):
  - Research Site, Harrow
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: No